CLINICAL TRIAL: NCT02034513
Title: A Randomised, Double Blind, Cross-over Trial Comparing the Safety and Efficacy of Insulin Degludec and Insulin Glargine, Both With Insulin Aspart as Mealtime Insulin in Subjects With Type 1 Diabetes (SWITCH 1)
Brief Title: A Trial Comparing the Safety and Efficacy of Insulin Degludec and Insulin Glargine, Both With Insulin Aspart as Mealtime Insulin in Subjects With Type 1 Diabetes
Acronym: SWITCH 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-3995; U1111-1129-9668 (Other: WHO); 2012-001930-32 (EudraCT Number)
Record Dates: First submitted 2014-01-07; First posted 2014-01-13 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg OD + IAsp followed by IGlar OD + IAsp (Experimental): Each treatment period consists of a 16-week wash-out period and a 16-week maintenance period
  Interventions: Drug: insulin degludec; Drug: insulin glargine; Drug: insulin aspart
- IGlar OD + IAsp followed by IDeg OD + IAsp (Active Comparator): Each treatment period consists of a 16-week wash-out period and a 16-week maintenance period
  Interventions: Drug: insulin degludec; Drug: insulin glargine; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Administered once daily, injected s.c. / subcutaneously (under the skin). Dose is individually adjusted.
Drug: insulin glargine — Administered once daily, injected s.c. / subcutaneously (under the skin). Dose is individually adjusted.
Drug: insulin aspart — Administered 2-4 times daily injected s.c. / subcutaneously (under the skin). Dose is individually adjusted.

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of the trial is to compare the safety and efficacy of insulin degludec (IDeg) and insulin glargine (IGlar), both with insulin aspart (IAsp) as mealtime insulin in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Subjects fulfilling at least one of the below criteria: a) Experienced at least one severe hypo episode within the last year (according to the ADA (American Diabetes Association) definition, April 2013) b) Moderate chronic renal failure, defined as glomerular filtration rate 30 - 59 mL/min/1.73 m^2 per CKD-Epi (chronic kidney disease epidemiology collaboration) c) Hypoglycaemic symptom unawareness d) Diabetes mellitus duration for more than 15 years e) Recent episode of hypoglycaemia (defined by symptoms of hypoglycaemia and/or episode with low glucose measurement (below or equal to 70 mg/dL [below or equal to 3.9 mmol/L])) within the last 12 weeks prior to Visit 1 (screening) - Male or female, age at least 18 years at the time of signing informed consent - Type 1 diabetes mellitus (diagnosed clinically) for at least 52 weeks prior to Visit 1 - Current treatment with a basal-bolus regimen consisting of neutral protamine Hagedorn (NPH) insulin OD (once daily) / BID (twice daily) or insulin detemir (IDet) OD / BID plus 2-4 daily injections of any rapid acting meal time insulin or CSII (with rapid acting insulin) for at least 26 weeks prior to Visit 1 - HbA1c (glycosylated haemoglobin) below or equal to 10% by central laboratory analysis - BMI (body mass index) below or equal to 45 kg/m^2 Exclusion Criteria: - Treatment with IGlar or IDeg within the last 26 weeks prior to Visit 1 (short term use [less than or equal to 2 weeks] is allowed, but not within 4 weeks prior to screening) - Use of any other anti-diabetic agent than those stated in the inclusion criteria within the last 26 weeks prior to Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2014-01-05 (Actual); Primary Completion 2016-01-11 (Actual); Study Completion 2016-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (90):
- United States (84):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Rancho Cucamonga, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Santa Monica, California
  - Novo Nordisk Investigational Site, Upland, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Cooper City, Florida
  - Novo Nordisk Investigational Site, Fleming Island, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Miami Springs, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Port Charlotte, Florida
  - Novo Nordisk Investigational Site, Port Orange, Florida
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Arlington Heights, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Crystal Lake, Illinois
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Anderson, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, West Des Moines, Iowa
  - Novo Nordisk Investigational Site, Lenexa, Kansas
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Livonia, Michigan
  - Novo Nordisk Investigational Site, Hazelwood, Missouri
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Hamilton, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Harrison, New York
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Jenkintown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Carrollton, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, El Paso, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Katy, Texas
  - Novo Nordisk Investigational Site, Mesquite, Texas
  - Novo Nordisk Investigational Site, Richardson, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Schertz, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Chesapeake, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Federal Way, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Richland, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Walla Walla, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Poland (5):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zabrze
- Novo Nordisk Investigational Site, Manatí, Puerto Rico

REFERENCES:
- [Result] Lane W, Bailey TS, Gerety G, Gumprecht J, Philis-Tsimikas A, Hansen CT, Nielsen TSS, Warren M; Group Information; SWITCH 1. Effect of Insulin Degludec vs Insulin Glargine U100 on Hypoglycemia in Patients With Type 1 Diabetes: The SWITCH 1 Randomized Clinical Trial. JAMA. 2017 Jul 4;318(1):33-44. doi: 10.1001/jama.2017.7115. PMID 28672316
- [Result] Evans M, Mehta R, Gundgaard J, Chubb B. Cost-Effectiveness of Insulin Degludec vs. Insulin Glargine U100 in Type 1 and Type 2 Diabetes Mellitus in a UK Setting. Diabetes Ther. 2018 Oct;9(5):1919-1930. doi: 10.1007/s13300-018-0478-1. Epub 2018 Aug 10. PMID 30097995
- [Result] DeVries JH, Bailey TS, Bhargava A, Gerety G, Gumprecht J, Heller S, Lane W, Wysham CH, Zinman B, Bak BA, Hachmann-Nielsen E, Philis-Tsimikas A. Day-to-day fasting self-monitored blood glucose variability is associated with risk of hypoglycaemia in insulin-treated patients with type 1 and type 2 diabetes: A post hoc analysis of the SWITCH Trials. Diabetes Obes Metab. 2019 Mar;21(3):622-630. doi: 10.1111/dom.13565. Epub 2018 Nov 26. PMID 30362250
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 90 sites in 2 countries, as follows: US: 84 sites, Poland: 6 sites.
Groups:
- Insulin Degludec/Insulin Glargine (IDeg/IGlar): Subjects received insulin degludec (IDeg) in treatment period 1 and insulin glargine (IGlar) in treatment period 2. Each treatment period consisted of a 16-week titration period and a 16-week maintenance period (total 32 weeks for each treatment period). IDeg and IGlar were administered subcutaneously (s.c.; under the skin) in the morning (from waking up to breakfast) or in the evening (from main evening meal to bedtime), as per randomisation and were to be taken once daily (OD) at the same time of day throughout the trial. To prevent an increased risk of hypoglycaemia in the first treatment month, the overall daily doses of IDeg and IGlar were reduced by 20% at the start of both the treatment periods. Doses of IDeg and IGlar were titrated individually. Titration of the dose was performed once weekly based on the lowest of 3 pre-breakfast self measured plasma glucose(SMPG) values measured on 3 consecutive days immediately prior to titration (fasting glycaemic target of 4.0-5.0 mmol/L)
- Insulin Glargine/Insulin Degludec (IGlar/IDeg): Subjects received IGlar in treatment period 1 and IDeg in treatment period 2. Each treatment period consisted of a 16-week titration period and a 16-week maintenance period (total 32 weeks for each treatment period). IGlar and IDeg were administered s.c. in the morning (from waking up to breakfast) or in the evening (from main evening meal to bedtime), as per randomisation and were to be taken OD at the same time of day throughout the trial. To prevent an increased risk of hypoglycaemia in the first treatment month, the overall daily doses of IGlar and IDeg were reduced by 20% at the start of both the treatment periods. Doses of IGlar and IDeg were titrated individually. Titration of the dose was performed once weekly based on the lowest of 3 pre-breakfast SMPG values measured on 3 consecutive days immediately prior to titration (fasting glycaemic target of 4.0-5.0 mmol/L).
Period: Overall Study
Arm/Group | Insulin Degludec/Insulin Glargine (IDeg/IGlar) | Insulin Glargine/Insulin Degludec (IGlar/IDeg)
Started | 249 | 252
Exposed | 249 | 251
Completed | 200 | 195
Not Completed | 49 | 57
Not completed — Adverse Event | 11 | 10
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 6 | 7
Not completed — Pregnancy | 0 | 3
Not completed — Protocol Violation | 7 | 10
Not completed — Withdrawal by Subject | 25 | 25
Not completed — Unclassified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline results are based on the full analysis set (FAS), which included all randomised subjects.
Groups:
- Insulin Degludec/Insulin Glargine (IDeg/IGlar): Subjects received IDeg in treatment period 1 and IGlar in treatment period 2. Each treatment period consisted of a 16-week titration period and a 16-week maintenance period (total 32 weeks for each treatment period). IDeg and IGlar were administered s.c.in the morning (from waking up to breakfast) or in the evening (from main evening meal to bedtime), as per randomisation and were to be taken OD at the same time of day throughout the trial. To prevent an increased risk of hypoglycaemia in the first treatment month, the overall daily doses of IDeg and IGlar were reduced by 20% at the start of both the treatment periods. Doses of IDeg and IGlar were titrated individually. Titration of the dose was performed once weekly based on the lowest of 3 pre-breakfast SMPG values measured on 3 consecutive days immediately prior to titration fasting glycaemic target of 4.0-5.0 mmol/L).
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Insulin Glargine (IDeg/IGlar) | Insulin Glargine/Insulin Degludec (IGlar/IDeg) | Total
Number analyzed (Participants) | 249 | 252 | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (13.7) | 46.4 (14.6) | 45.9 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 109 | 232
  Male | 126 | 143 | 269
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — Population: The number of subjects that contributed to the measurement of HbA1c
  Percentage of HbA1c
    number analyzed (Participants) | 248 | 252 | 500
    (all) | 7.7 (1.0) | 7.5 (1.0) | 7.6 (1.0)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Population: The number of subjects that contributed to the measurement of FPG
  mg/dL
    number analyzed (Participants) | 248 | 252 | 500
    (all) | 165.1 (77.3) | 174.4 (81.7) | 169.8 (79.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Severe or BG (Blood Glucose) Confirmed Symptomatic Hypoglycaemic Episodes During the Maintenance Period
Description: Severe or blood glucose (BG) confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe and/or BG confirmed by a plasma glucose value of <3.1 mmol/L (56 mg/dL), with symptoms consistent with hypoglycaemia. Treatment emergent hypoglycaemic episode was defined as an event with onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment. Maintenance period: 16 weeks of treatment, in each treatment period (Week 16-32 and Week 48-64).
Time Frame: A 16-week treatment period.
Population: The trial followed a cross over design. Descriptive analysis was based on the safety analysis set (SAS: subjects receiving at least 1 dose of the investigational product, IDeg or its comparator, IGlar). Number of subjects analysed=subjects in the SAS, who were exposed in at least one maintenance period.
Measure: Number; unit: Event
Groups:
- Insulin Degludec (IDeg): Subjects received IDeg in treatment period 1 (from treatment sequence IDeg/IGlar) and in treatment period 2 (from treatment sequence IGlar/IDeg). Each treatment period consisted of a 16-week titration period and a 16-week maintenance period (total 32 weeks for each treatment period). IDeg was administered s.c. in the morning (from waking up to breakfast) or in the evening (from main evening meal to bedtime), as per randomisation and was to be taken OD at the same time of day throughout the trial. To prevent an increased risk of hypoglycaemia in the first treatment month, the overall daily doses of IDeg were reduced by 20% at the start of both the treatment periods. Doses of IDeg were titrated individually. Titration of the dose was performed once weekly based on the lowest of 3 pre-breakfast SMPG values measured on 3 consecutive days immediately prior to titration (fasting glycaemic target of 4.0-5.0 mmol/L).
- Insulin Glargine (IGlar): Subjects received IGlar in treatment period 1 (from treatment sequence IGlar/IDeg) and in treatment period 2 (from treatment sequence IDeg/IGlar). Each treatment period consisted of a 16-week titration period and a 16-week maintenance period (total 32 weeks for each treatment period). IGlar was administered s.c. in the morning (from waking up to breakfast) or in the evening (from main evening meal to bedtime), as per randomisation and was to be taken OD at the same time of day throughout the trial. To prevent an increased risk of hypoglycaemia in the first treatment month, the overall daily doses of IGlar were reduced by 20% at the start of both the treatment periods. Doses of IGlar were titrated individually. Titration of the dose was performed once weekly based on the lowest of 3 pre-breakfast SMPG values measured on 3 consecutive days immediately prior to titration (fasting glycaemic target of 4.0-5.0 mmol/L).
Arm/Group | Insulin Degludec (IDeg) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 418 | 422
Event | 2772 | 3126
Statistical Analysis 1: Comparison: Insulin Degludec (IDeg) vs Insulin Glargine (IGlar); Statistical analysis was performed on the FAS. Number of subjects analysed=subjects in the FAS, who were exposed in at least one maintenance period. Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 1: Number of treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the maintenance period; Test type: Non-Inferiority or Equivalence — Non-inferiority was considered confirmed if the 95% confidence interval for the rate ratio (IDeg/IGlar) was ≤1.10 or equivalently if the p-value for the 1-sided test of H0: RR >1.10 against HA: RR ≤1.10 was less than 2.5%, where RR is the estimated rate ratio IDeg/IGlar; p < 0.0001, Poisson; Treatment ratio = 0.89, 95% CI 2-sided [0.85 to 0.94] — If non-inferiority was confirmed the superiority of IDeg/IGlar was investigated outside of the test hierarchy. Superiority was considered confirmed if the upper bound of the 2-sided 95% confidence interval was <1.00

2. Secondary Outcome: Number of Treatment Emergent Severe or BG Confirmed Symptomatic Nocturnal Hypoglycaemic Episodes During the Maintenance Period
Description: Severe or BG confirmed symptomatic nocturnal hypoglycaemic episodes were defined as episodes that were severe and/or BG confirmed by a plasma glucose value of <3.1 mmol/L (56 mg/dL), with symptoms consistent with hypoglycaemia and with time of onset between 00:01 and 05.59 a.m., both inclusive. Treatment emergent hypoglycaemic episode was defined as an event with onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment.
Time Frame: After 16 weeks of treatment, in each treatment period (Week 16-32 and Week 48-64)
Population: The trial followed a cross over design. Descriptive analysis was based on the SAS. Number of subjects analysed=subjects in the SAS, who were exposed in at least one maintenance period.
Measure: Number; unit: Event
Arm/Group | Insulin Degludec (IDeg) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 418 | 422
Event | 349 | 544
Statistical Analysis 1: Comparison: Insulin Degludec (IDeg) vs Insulin Glargine (IGlar); Statistical analysis was performed on the FAS. Number of subjects analysed=subjects in the FAS, who were exposed in at least one maintenance period. Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 2: Number of treatment-emergent severe or BG confirmed symptomatic nocturnal hypoglycaemic episodes during the maintenance period; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, Poisson; Treatment ratio = 0.64, 95% CI 2-sided [0.56 to 0.73] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Proportion of Subjects With One or More Severe Hypoglycaemic Episodes During the Maintenance Period
Description: Percentage of subjects who experienced one or more severe hypoglycaemic episodes during the maintenance period. Severe hypoglycaemia (according to the American Diabetes Association 2013 definition): A hypoglycaemic episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose values may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: After 16 weeks of treatment, in each treatment period (Week 16-32 and Week 48-64)
Population: as for outcome 2
Measure: Number; unit: Percentage of subjects
Arm/Group | Insulin Degludec (IDeg) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 418 | 422
Percentage of subjects | 10.3 | 17.1
Statistical Analysis 1: Comparison: Insulin Degludec (IDeg) vs Insulin Glargine (IGlar); Statistical analysis was performed on the FAS. Number of subjects analysed=subjects in the FAS, who were exposed in both the maintenance periods. Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 3: Proportion of subjects with one or more severe hypoglycaemic episodes during the maintenance period; Test type: Superiority or Other; p = 0.0016, McNemar — Superiority was confirmed if the p-value was less than 0.025

4. Secondary Outcome: Incidence of Treatment Emergent Adverse Events
Description: Treatment emergent adverse event was defined as an event with onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment.
Time Frame: During 32 weeks of treatment for each treatment period
Population: The trial followed a cross over design. Results are based on the SAS.
Measure: Number; unit: Event
Arm/Group | Insulin Degludec (IDeg) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 454 | 460
Event | 925 | 937

5. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline in HbA1c (glycosylated haemoglobin) at week 32 (treatment period 1) and at week 64 (treatment period 2). Week 32 HbA1c absolute value was considered as baseline for calculating change from baseline in HbA1c at week 64.
Time Frame: Week 32, Week 64
Population: Both descriptive analysis and statistical analysis were based on the FAS. Here, 'n' specifies the number of subjects with available data at specified time-point.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Insulin Degludec/Insulin Glargine (IDeg/IGlar) | Insulin Glargine/Insulin Degludec (IGlar/IDeg)
Number analyzed (Participants) | 249 | 252
Percentage of glycosylated haemoglobin
  week 32 (n=209, 205) | -0.73 (0.89) | -0.66 (0.76)
  week 64 (n=203, 199) | 0.04 (0.51) | 0.17 (0.64)
Statistical Analysis 1: Comparison: Insulin Degludec/Insulin Glargine (IDeg/IGlar) vs Insulin Glargine/Insulin Degludec (IGlar/IDeg); Change from baseline in HbA1c at week 32 (treatment period 1). Before testing the primary endpoint, the secondary supportive efficacy endpoint "Change from baseline in HbA1c after 32 weeks of treatment" was tested for non-inferiority as a prerequisite for testing the primary endpoint. Analysis was based on mixed model for repeated measurement (MMRM); treatment, sex, region, pre-trial insulin treatment regimen, visit and dosing time were fixed effects, and age and baseline HbA1c were covariates; Test type: Non-Inferiority or Equivalence — Non-inferiority was considered confirmed if the upper bound of the two-sided 95% confidence interval was below or equal to 0.40%. Comparison groups: IDeg versus IGlar. Number of subjects included in analysis is 437 (n=220 for IDeg and n=217 for IGlar); Treatment contrast = 0.03, 95% CI 2-sided [-0.10 to 0.15]
Statistical Analysis 2: Comparison: Insulin Degludec/Insulin Glargine (IDeg/IGlar) vs Insulin Glargine/Insulin Degludec (IGlar/IDeg); Change from baseline in HbA1c at week 64 (treatment period 2). The baseline values are week 32 values. Before the primary endpoint was tested, the secondary supportive efficacy endpoint "Change from baseline in HbA1c after 32 weeks of treatment" was tested for non-inferiority as prerequisite for testing the primary endpoint. Analysis was based on MMRM; treatment, sex, region, pre-trial insulin treatment regimen, visit and dosing time were fixed effects, and age and baseline HbA1c were covariates; Test type: Non-Inferiority or Equivalence — Non-inferiority was considered confirmed if the upper bound of the two-sided 95% confidence interval was below or equal to 0.40%. Comparison groups: IDeg versus IGlar. Number of subjects included in analysis is 410 (n=202 for IDeg and n=208 for IGlar); Treatment contrast = 0.11, 95% CI 2-sided [-0.00 to 0.23]

6. Secondary Outcome: FPG (Fasting Plasma Glucose)
Description: Fasting plasma glucose values at week 32 and week 64.
Time Frame: Week 32 and Week 64
Population: Results are based on the FAS. Here, 'n' specifies the number of subjects with available data at specified time-point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Insulin Glargine (IDeg/IGlar) | Insulin Glargine/Insulin Degludec (IGlar/IDeg)
Number analyzed (Participants) | 249 | 252
mmol/L
  week 32 (n=208, 204) | 7.45 (3.57) | 8.12 (3.56)
  week 64 (n=203, 201) | 8.62 (4.24) | 7.54 (3.68)

ADVERSE EVENTS:
Time Frame: From the first day of exposure to randomised treatment and no later than the last day of randomised treatment (64 weeks).
Description: Subjects in the SAS contributed to the evaluation of adverse events. The following displayed "number of subjects at risk"=454 and 460 for IDeg and IGlar, respectively (i.e, out of a total of 500 exposed subjects, 454 received IDeg and 460 received IGlar in a cross-over manner in 2 treatment periods.
Arm/Group | Insulin Degludec (IDeg) | Insulin Glargine (IGlar)
Serious Adverse Events (participants affected / at risk) | 58/454 | 70/460
Other Adverse Events (participants affected / at risk) | 97/454 | 97/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec (IDeg) (N=454) | Insulin Glargine (IGlar) (N=460)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (4) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 17 (32) | 33 (47)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 3 (5) | 5 (5)
Hypoglycaemic unconsciousness (Nervous system disorders) | 18 (23) | 19 (24)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pancreas transplant (Surgical and medical procedures) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec (IDeg) (N=454) | Insulin Glargine (IGlar) (N=460)
Nasopharyngitis (Infections and infestations) | 68 (92) | 61 (73)
Upper respiratory tract infection (Infections and infestations) | 29 (34) | 39 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.